CLINICAL TRIAL: NCT00863031
Title: A Randomised Controlled Trail on the Effectiveness of Screening and Brief Counselling (Problem-Solving Therapy) for Elderly Patients With Psychological Problems in Primary Care.
Brief Title: A Trial on the Effectiveness of Screening and Brief Problem-Solving Therapy (PST) for Elderly Patients With Psychological Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health Care and Promotion Fund, Government of the Hong Kong SAR (Unknown)
Responsible Party: Cindy L.K. Lam, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKCTR-497
Record Dates: First submitted 2009-03-15; First posted 2009-03-17 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Undiagnosed Psychological Problems
Keywords: mental health; problem-solving therapy; elderly; health-related quality of life; primary care; Chinese
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- problem-solving therapy (Experimental): Three sessions of brief problem-solving counselling at week 1, 3 and 5 by a family doctor.
  Interventions: Behavioral: problem-solving therapy
- viewing video (Placebo Comparator): Three sessions of health education viewing video in groups of 3 to 5 people
  Interventions: Behavioral: Video-viewing

INTERVENTIONS:
Behavioral: problem-solving therapy — Three sessions of problem-solving therapy at week 1, 3 and 5.
  Arms: problem-solving therapy
Behavioral: Video-viewing — Three sessions of viewing health educational videos.
  Arms: viewing video

SUMMARY:
The aim of this study was to determine whether screening followed by brief PSC provided by primary care doctors could improve the quality of life of elderly patients with unrecognized psychological problems in primary care. The following hypotheses were tested:

1. Elderly patients screened positive of psychological problems had poorer health-related quality of life (HRQOL) than those who were screened negative.
2. Primary care doctors could be trained to provide brief PST.
3. Brief PST by a trained primary care doctor could improve the HRQOL of the elderly who were screened positive for psychological problems.

DETAILED DESCRIPTION:
Design & methods: A prospective single-blind randomised controlled trial (RCT) on 299 patients aged 60 or above without any known psychological diseases but screened positive for psychological problems by the Hospital Anxiety and Depression Scale (HADS). Subjects were randomised to problem-solving (PST) or video-viewing (placebo). All subjects continued with their usual care and were followed up by telephone at 6, 12, 26 and 52 weeks.Changes in SF-36 HRQOL scores, HADS scores and monthly consultation rates at 6, 12, 26 and 52 weeks within groups and between groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 or above
* not known to have any psychological problem
* HADS Depression score 6 or above, or Anxiety Score 3 or above
* Written consent to study

Exclusion Criteria:

* known psychological disease diagnosed by a registered doctor
* history of taking any psychotropic drug prescribed by a registered doctor within the last year;
* suicidal plan or strong suicidal thought;
* psychotic symptom;
* impairment in cognitive function; or
* communication problem.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2002-11; Primary Completion 2005-12 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life scores | 6, 12, 26 and 52 weeks

SECONDARY OUTCOMES:
Hospital Anxiety & Depression Scale scores | 6, 12, 26 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, MD, Principal Investigator — Family Medicine Unit, Faculty of Medicine, HKU
Locations (1):
- Two General Outpatient Clinics, Hong Kong, Hong Kong

REFERENCES:
- [Result] Lam C.L.K., Lee P.W.H., Fong D.Y.T. and Lam T.P., A randomised controlled trial on the effectiveness of screening and brief problem-solving counselling for elderly patients with undiagnosed psychological problems in primary care., Hong Kong Medical Journal. HK Academy of Medicine Press, 2008, 14: 31-35.